CLINICAL TRIAL: NCT05435950
Title: Prospective, Monocenter, Non-randomized Clinical Investigation Evaluating the Safety, Clinical Performance and Effectiveness of Sono-instruments for the Percutaneous Ultrasound-guided Treatment of Carpal Tunnel Syndrome and Trigger Finger
Brief Title: Clinical Investigation on Safety, Performance and Effectiveness of Sono-instruments
Acronym: SONO-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spirecut (Industry)
Collaborators: Archer Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SONO-01
Record Dates: First submitted 2022-06-09; First posted 2022-06-28 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Trigger Finger; Trigger Thumb; Carpal Tunnel Syndrome
MeSH Terms: conditions — Trigger Finger Disorder; Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult participants with Carpal Tunnel syndrome or with Trigger Finger/Thumb (Experimental)
  Interventions: Device: Sono-Intruments

INTERVENTIONS:
Device: Sono-Intruments — Spirecut's single use, pre-CE Sono-Instruments (SI) allow the percutaneous treatment of Carpal Tunnel (CT) syndrome and Trigger Finger/thumb (TF) under sonography (instead of open or endoscopic approach).
  Two models will be assessed:
  * The Carpal Tunnel Sono-Instrument® (CT-SI), for CT syndrome release, by progressively cutting the transverse carpal ligament.
  * The Trigger Finger Sono-Instrument® (TF-SI), for TF release by progressively cutting the A1 annual pulley.

SUMMARY:
Carpal Tunnel (CT) syndrome is a collection of characteristic symptoms and signs that occurs following compression of the median nerve within the CT. In Trigger Finger / trigger thumb (TF), one of the most common causes of hand pain and disability, the flexor tendon causes painful popping or snapping as the patient flexes and extends the digit. In case of failure of non-operative treatments, patients with CT syndrome or TF are operated. Clearly any improvement in surgical device design would be of great advantage to the patient and the surgeon. Spirecut's single use, pre-CE Sono-Instruments (SI) allow the percutaneous treatment of Carpal Tunnel (CT)syndrome and Trigger Finger/thumb (TF) under sonography (instead of open or endoscopic approach). Two models will be assessed in this clinical investigation:

1. The Carpal Tunnel Sono-Instrument® (CT-SI), for CT syndrome release, by progressively cutting the transverse carpal ligament.
2. The Trigger Finger Sono-Instrument® (TF-SI), for TF release by progressively cutting the A1 annual pulley.

Using those SI, surgical procedures can be performed without endangering adjacent structures (e.g. median nerve and branches, ulnar pedicle, superficial carpal arch, digital pedicles, flexor tendons).

ELIGIBILITY:
Participants with Carpal tunnel syndrome:

Inclusion Criteria:

* Adults ≥ 18 years of age;
* Primary CT confirmed by typical symptoms, signs and altered nerve conduction studies;
* Pain and/or numbness in the hand which worsen at night (or are present only at night);
* Participant and investigator signed and dated the Informed Consent Form (ICF) prior to the index-procedure.

Participants with Trigger Finger/thumb:

Inclusion Criteria:

* Adults ≥ 18 years of age;
* Typical signs and symptoms of TF/thumb caused by friction or blockade of flexor tendon(s) in digital sheath, without flexion contracture over 30° of the proximal interphalangeal (or interphalangeal for the thumb) joint, confirmed by altered flexor tendon(s) gliding and/or increased thickness of A1 digital pulley under sonography (sonography can be done just before the operation, that is after signature of the ICF);
* Participant and investigator signed and dated the ICF prior to the index-procedure.

Exclusion criteria:

Participants with one or more of the following conditions are excluded from the study:

* Dwarfism or participants with small size hand/CT/TF-thumb;
* Past or active infection;
* Known allergic reaction to metals;
* Coagulation problems, with significant risk of per/postoperative bleeding;
* In case of TF: long evolution, with ankylosis of the proximal interphalangeal joint;
* In case of CT: severe median nerve dysfunction;
* Previous facture or dislocation in the operated area or any affection causing malalignment or distortion of the local skeleton due to trauma, arthritis or other causes;
* Other known clinical risks outweighing the expected clinical benefits or increasing the risk of a postoperative lesion (e.g. tissue adhesions, anatomical abnormalities, neuro-vascular structures in the zone of the intended release, local tumors);
* Insufficient sonographic identification of the operated tissue;
* Previous attempt to treat the condition;
* Currently receiving treatment for CT or TF;
* Contra-indication to local anesthesia (general, regional or local);
* Participant unable (vulnerable participant)/unwilling to provide informed consent;
* Participant is enrolled in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Safety of percutaneous surgery performed with Sono-Instuments | During the index procedure
  Number of peri- and post-operative (serious) adverse events, including operative and post-operative complications (e.g. infection), symptomatic recurrences and re-interventions.
Safety of percutaneous surgery performed with Sono-Instuments | Within 1 week after the procedure
  Number of peri- and post-operative (serious) adverse events, including operative and post-operative complications (e.g. infection), symptomatic recurrences and re-interventions.
Safety of percutaneous surgery performed with Sono-Instuments | 6 weeks after the procedure
  Number of peri- and post-operative (serious) adverse events, including operative and post-operative complications (e.g. infection), symptomatic recurrences and re-interventions.

SECONDARY OUTCOMES:
Performance of Sono-Instruments during percutaneous surgery | During the index procedure
  Ease of positioning of Sono-Instruments during percutaneous surgery. A score ranging from 0 (very unsatisfied) to 4 (very satisfied) will be documented by surgeons experienced in performing percutaneous surgery.
Performance of Sono-Instruments during percutaneous surgery | During the index procedure
  Maneuverability of Sono-Instruments during percutaneous surgery. A score ranging from 0 (very unsatisfied) to 4 (very satisfied) will be documented by surgeons experienced in performing percutaneous surgery.
Performance of Sono-Instruments during percutaneous surgery | During the index procedure
  Visibility (location and orientation) of the Sono-Instruments under sonography. A score ranging from 0 (very unsatisfied) to 4 (very satisfied) will be documented by surgeons experienced in performing percutaneous surgery.
Performance of Sono-Instruments during percutaneous surgery | During the index procedure
  Technical success of the surgical procedure, defined as percutaneous surgery as intended without technical difficulties and without conversion to another surgical intervention.
Pre-operative pain | During screening
  Pain is assessed using the Numeric pain Rating Scale (NRS) in rest and activity (e.g. use for light daily activities like eating with the operated hand, putting the clothes on, washing the hands etc.). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Post-operative pain of percutaneous surgery performed with Sono-Instruments | Within 1 week after the procedure
  Pain is assessed using the Numeric pain Rating Scale (NRS) in rest and activity (e.g. use for light daily activities like eating with the operated hand, putting the clothes on, washing the hands etc.). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Post-operative pain of percutaneous surgery performed with Sono-Instruments | 6 weeks after the procedure
  Pain is assessed using the Numeric pain Rating Scale (NRS) in rest and activity (e.g. use for light daily activities like eating with the operated hand, putting the clothes on, washing the hands etc.). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | During screening
  Document use of anti-inflammatory/pain medications.
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | During screening
  Document what the participant cannot do with his/her affected hand.
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | During screening
  Quick Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire, including 11 items with 5 response options each (1 = no problem with activity, 5 = activity is not possible).
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | During screening
  Boston Carpal Tunnel Questionnaire Symptom Severity (BCTQ-SS) in patients with carpal tunnel syndrome, including 11 items with 5 response options each (1 = low level of symptoms/difficulty, 5 = highly symptomatic/unable to complete functional tasks).
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | During screening
  Boston Carpal Tunnel Questionnaire Functional Scale (BCTQ-FS) in patients with carpal tunnel syndrome, including 8 items with 5 response options each (1 = low level of symptoms/difficulty, 5 = highly symptomatic/unable to complete functional tasks).
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | During screening
  Noting of numbness/pain at night in patients with carpal tunnel syndrome.
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | During screening
  Quinnell grading system in patients with trigger finger/thumb, including 2 items with 5 response options each (0 = normal movement of the digit, 4 = fixed deformity).
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | Within 1 week after the procedure
  Document use of anti-inflammatory/pain medication.
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | 6 weeks after the procedure
  Document use of anti-inflammatory/pain medication.
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | Within 1 week after the procedure
  Document what the participant cannot do with his/her affected hand.
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | 6 weeks after the procedure
  Document what the participant cannot do with his/her affected hand.
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | Within 1 week after the procedure
  Quick Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire, including 11 items with 5 response options each (1 = no problem with activity, 5 = activity is not possible).
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | 6 weeks after the procedure
  Quick Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire, including 11 items with 5 response options each (1 = no problem with activity, 5 = activity is not possible).
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | Within 1 week after the procedure
  Post-operative time to return to activities of daily living as prescribed by the doctor and effectively done by participant.
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | Within 1 week after the procedure
  Post-operative time to return to work as prescribed by the doctor and effective return to work for participants that are employed.
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | Within 1 week after the procedure
  Number of days between surgery and washing of the operated hand for the first time.
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | Within 1 week after the procedure
  Boston Carpal Tunnel Questionnaire Symptom Severity (BCTQ-SS) in patients with carpal tunnel syndrome, including 11 items with 5 response options each (1 = low level of symptoms/difficulty, 5 = highly symptomatic/unable to complete functional tasks).
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | 6 weeks after the procedure
  Boston Carpal Tunnel Questionnaire Symptom Severity (BCTQ-SS) in patients with carpal tunnel syndrome, including 11 items with 5 response options each (1 = low level of symptoms/difficulty, 5 = highly symptomatic/unable to complete functional tasks).
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | Within 1 week after the procedure
  Boston Carpal Tunnel Questionnaire Functional Scale (BCTQ-FS) in patients with carpal tunnel syndrome, including 8 items with 5 response options each (1 = low level of symptoms/difficulty, 5 = highly symptomatic/unable to complete functional tasks).
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | 6 weeks after the procedure
  Boston Carpal Tunnel Questionnaire Functional Scale (BCTQ-FS) in patients with carpal tunnel syndrome, including 8 items with 5 response options each (1 = low level of symptoms/difficulty, 5 = highly symptomatic/unable to complete functional tasks).
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | Within 1 week after the procedure
  Noting of numbness/pain at night in patients with Carpal Tunnel Syndrome.
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | 6 weeks after the procedure
  Noting of numbness/pain at night in patients with Carpal Tunnel Syndrome.
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | Within 1 week after the procedure
  Noting of pillar pain in patients with Carpal Tunnel Syndrome.
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | 6 weeks after the procedure
  Noting of pillar pain in patients with Carpal Tunnel Syndrome.
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | Within 1 week after the procedure
  Quinnell grading system in patients with trigger finger/thumb, including 2 items with 5 response options each (0 = normal movement of the digit, 4 = fixed deformity).
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | 6 weeks after the procedure
  Quinnell grading system in patients with trigger finger/thumb, including 2 items with 5 response options each (0 = normal movement of the digit, 4 = fixed deformity).
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | Within 1 week after the procedure
  Modified Patel and Bassini's grading system in patients with trigger finger/thumb, including 2 items with 4 response options each (1 = no improvement, 4 = full improvement).
Clinical effectiveness of percutaneous surgery performed with Sono-Instruments | 6 weeks after the procedure
  Modified Patel and Bassini's grading system in patients with trigger finger/thumb, including 2 items with 4 response options each (1 = no improvement, 4 = full improvement).

CONTACTS AND LOCATIONS:
Locations (1):
- Erasme University Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No